CLINICAL TRIAL: NCT06145763
Title: Digital Smoking Cessation Intervention for Nationally-Recruited American Indians and Alaska Natives: A Full-Scale Randomized Controlled Trial (IndigeQuit)
Brief Title: A Digital Smoking Cessation Intervention for Helping American Indians and Alaska Natives Quit Smoking, IndigeQuit Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RG1123796; NCI-2023-09049 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20279 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA284687 (NIH)
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Specimen Handling; Smoking Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Random assignments will be concealed from participants and research staff throughout the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (IndigeQuit app) (Experimental): Participants use the IndigeQuit app, which includes setting up a personalized quit plan, participating in eight levels of the content, receiving on-demand help in coping with smoking urges, and tracking their daily smoking behaviors for at least 45 days on study.
  Interventions: Procedure: Biospecimen Collection; Behavioral: Smoking Cessation Intervention; Other: Survey Administration
- Arm II (NCI QuitGuide app) (Active Comparator): Participants use the NCI QuitGuide app for at least 45 days on study.
  Interventions: Procedure: Biospecimen Collection; Behavioral: Smoking Cessation Intervention; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Ancillary studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Behavioral: Smoking Cessation Intervention — Use IndigeQuit smartphone app
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: Arm I (IndigeQuit app)
Behavioral: Smoking Cessation Intervention — Use NCI QuitGuide smartphone app
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: Arm II (NCI QuitGuide app)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial compares a new smoking cessation smartphone application (app) (IndigeQuit) to an existing smarphone app (National Cancer Institute [NCI] QuitGuide) for helping American Indians and Alaska Natives (AI/ANs) quit smoking. Compared to other racial/ethnic groups, AIANs have 6 times higher rates of developing smoking-related cancers, including lung cancer. Commercial cigarette smoking accounts for half of all deaths among AIANs nationwide. AIANs' often lack of access to smoking cessation interventions, which may be due to inequities in the healthcare system, lack of health insurance, living in rural areas, systemic racism, and historical trauma. There is also a lack of effective smoking cessation interventions for AIANs. Smartphone apps have the potential to deliver a low-cost smoking cessation intervention with wide reach to AIANs. Apps require no in-person delivery and no provider training, do not require integration into complex hospital systems, can be freely accessed on an app store, and are available at any time and any place. IndigeQuit is a behavioral intervention designed to help adults stop smoking by teaching skills for coping with smoking urges, staying motivated, and preventing relapse. The IndigeQuit app intervention may be more effective than the currently available NCI QuitGuide app at helping AIANs quit smoking.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants use the IndigeQuit app, which includes setting up a personalized quit plan, participating in eight levels of the content, receiving on-demand help in coping with smoking urges, and tracking their daily smoking behaviors for at least 45 days on study.

ARM II: Participants use the NCI QuitGuide app for at least 45 days on study.

After completion of study intervention, patients are followed up at 3, 6, and 12-months.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as American Indian or Alaska Native, either alone or in combination with other races
* Age 18 and older
* Has smoked daily for the past year
* Interest in quitting smoking within the next 30 days
* Willing to be randomly assigned to either app
* Have daily access to their own Android or iPhone
* Able to download a smartphone app
* Be willing and able to read English
* Not currently or within past 30 days using other smoking cessation behavioral interventions or smoking cessation pharmacotherapies
* Have never participated in our prior research
* Have no other household or family member participating
* Being willing to complete the 3, 6, and 12-month follow-up assessments
* Providing email, phone number(s), and mailing address
* Living off United States (US) AI/AN tribal reservations or living on five Northern Plains tribal reservations from whom we would obtain approvals to recruit

Exclusion Criteria:

* Currently (i.e., within past 30 days) using other smoking cessation behavioral interventions
* Has participated in our prior research trials
* Has used the National Cancer Institute's (NCI's) QuitGuide app
* Not willing to complete a follow-up survey at 3, 6, and 12 months post-randomization
* Not providing email, phone number(s), and mailing address

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 776 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
30-day point prevalence abstinence (PPA) | At 12 months post randomization
  Will be assessed based on self-report with biochemical verification of salivary cotinine. For each comparison of treatment arms on cessation outcomes, will use a logistic regression model.

SECONDARY OUTCOMES:
30-day PPA | At 3- and 6-months post randomization
  Will be assessed based on self-report with biochemical verification of salivary cotinine. For each comparison of treatment arms on cessation outcomes, will use a logistic regression model.
Self-reported 24-hour PPA | At the 3, 6, and 12-month follow-ups
  A secondary definition of cessation will include self-reported abstinence from cigarettes and all other commercial nicotine-containing tobacco products (i.e., e-cigarettes or vaping, chewing tobacco, snus, hookahs, cigars, cigarillos, tobacco pipes, kreteks). Will be assessed based on self-report with biochemical verification of salivary cotinine. For each comparison of treatment arms on cessation outcomes, will use a logistic regression model.
Self-reported 7-day PPA | At the 3, 6, and 12-month follow-ups
  A secondary definition of cessation will include self-reported abstinence from cigarettes and all other commercial nicotine-containing tobacco products (i.e., e-cigarettes or vaping, chewing tobacco, snus, hookahs, cigars, cigarillos, tobacco pipes, kreteks). Will be assessed based on self-report with biochemical verification of salivary cotinine. For each comparison of treatment arms on cessation outcomes, will use a logistic regression model.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B. Bricker, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No